CLINICAL TRIAL: NCT01349088
Title: Phase I/II Trial of Motesanib in Combination With Ixabepilone and Capecitabine in Women With Locally Recurrent or Metastatic Breast Cancer
Brief Title: Investigational Drug in Combination With Two Chemotherapy Drugs in Women With Locally Recurrent or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other); Amgen (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10G.30; 2009-34 (Other: CCRRC); JT 1502 (Other: JeffTrial Number)
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Stage IV Breast Cancer
Keywords: breast cancer; metastatic breast cancer; stage IV breast cancer; motesanib; ixabepilone; capecitabine
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Capecitabine; motesanib diphosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Motesanib (Experimental): Eligible patients will be enrolled to receive ixabepilone, capecitabine, plus motesanib.
  Interventions: Drug: Ixabepilone; Drug: Capecitabine; Drug: Motesanib

INTERVENTIONS:
Drug: Ixabepilone — Patients will receive ixabepilone at 40 mg/m2.
  Other Names: azaepothilone B; BMS-247550
Drug: Capecitabine — Patients will receive capecitabine at 2000 mg/m2.
  Other Names: Xeloda
Drug: Motesanib — Patient will receive motesanib at 100mg or 125mg once daily dependent on outcome of Phase I, which will involve the first 3-6 patients.
  Other Names: Motesanib diphosphate; AMG 706

SUMMARY:
In 2008 there were more than 40,000 deaths caused by metastatic breast cancer in the United States. The development of new treatment strategies is essential to improve outcome for patients with metastatic breast cancer

There is significant preclinical and clinical evidence indicating that creating new blood vessels (neoangiogenesis) to provide nutrients to solid tumors, including breast cancer, provides the necessary conditions to allow tumor growth. Vascular endothelial growth factor (VEGF) is one of the important molecules regulating new blood vessel formations and subsequent invasion and metastases. As a result, agents that inhibit VEGF are of substantial interest for the treatment of advanced diseases.

This study will further the body of research of motesanib which has been shown in preclinical pharmacology and clinical pharmacology studies to be a potent, orally bioavailable multi-kinase inhibitor with anti-angiogenic and anti-tumor activity achieved by selectively targeting all known VEGF, platelet-derived growth factor (PDGF), and Kit receptors.

DETAILED DESCRIPTION:
Endocrine therapy and chemotherapy (using either sequential single agents or combination regimens) remain the principal treatments for women with metastatic breast cancer. A wide variety of classes of chemotherapeutic agents have demonstrated anti-tumor activity as single agents or in combination regimens. Cytotoxic chemotherapeutic agents have been the mainstay of cancer therapies for many years and have improved survival in many disease settings. Median survivals remain approximately two years for women with metastatic breast cancer, and less than 3% of patients experience long-term survival after initiation of treatment. The development of new treatment strategies is therefore essential to improve outcome for patients with metastatic breast cancer.

One of the most promising pathways for the development of new anti-neoplastic agents is targeting tumor vascular endothelium. There is significant preclinical and clinical evidence indicating that tumor neoangiogenesis is critical in pathogenesis and progression of solid tumors, including breast cancer. Of the numerous known growth factors that have been implicated in tumor angiogenesis, vascular endothelial growth factor (VEGF) is one of the important molecules regulating new blood vessel formations and subsequent invasion and metastases. As a result, agents that inhibit VEGF are of substantial interest for the treatment of advanced diseases. More thorough elucidation of mechanisms behind intrinsic and acquired resistance therefore is imperative disease and to identify patients most likely to benefit from treatment options.

Motesanib has been shown in preclinical pharmacology and PK studies to be a potent, orally bioavailable multi-kinase inhibitor with anti-angiogenic and anti-tumor activity achieved by selectively targeting all known VEGF, PDGF and Kit receptors. It has an acceptable safety profile in both non-clinical and clinical studies, and a PK profile that appears suitable for daily oral dosing in humans.

The investigational product motesanib (Amgen) is a small molecule tyrosine kinase inhibitor with high efficacy against VEGFR and c-Kit kinases. C-kit has been detected in 12% of breast cancers, correlating with basal or triple-negative breast cancer. In addition, efficacy of the drug has been noted to PDGFRα, which is expressed in approximately 40% of breast cancers and is associated with aggressive disease, metastatic invasion and poor prognosis. Importantly, in more than half (56%) of these cases, the carcinoma cells bearing the receptors expressed the PDGF-A ligand, suggesting an autocrine loop and a cancer cell-autonomous process. Cancer cell-autonomous pathways are especially attractive as drug targets against metastatic breast cancer because they are expected to continue to be functional at metastatic sites, since they do not depend on stromal factors.

The primary molecular target of motesanib, VEGFR, is intriguing because neovascularization is expected to be required also at metastatic sites. A preliminary analysis revealed that VEGF expression correlated with the triple-negative, basal breast cancer subtype and poor outcome. Importantly, PDGF receptors are also present on vascular pericytes, cells required for adequate vascularization. Thus, motesanib is a unique multikinase inhibitor that targets both growth factor receptors on the carcinoma cells and growth factor receptors related to neovascularization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast regardless of ER, PR and Her2 status with locally recurrent or metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* Disease progression after at least 1, but no more than 2, prior chemotherapy regimens for metastatic disease.
* Patients with hormone-sensitive tumors must have received prior hormonal therapy and not be amenable to further hormonal therapy.
* Patients with HER2/neu-overexpressing tumors (3+ by immunohistochemistry or amplified by fluorescent in situ hybridization) should have received trastuzumab (Herceptin®) and/or lapatinib (Tykerb®) in the adjuvant or metastatic setting (unless contraindicated) and have progressed while on treatment of metastatic disease or within 12 months of completion of adjuvant therapy.
* Patients will eligible if they have tumors that express one of the motesanib-directed tyrosine kinase markers, the target markers:(PDGFR, VEGFR, c-Kit) as determined by study pathologist. Immunohistochemical assays for these markers are provided by grant consortium partner and CLIA-certified diagnostics laboratory MDRG.
* Measurable disease per RECIST (Response Evaluation Criteria in Solid Tumor) guidelines.
* Complete radiology and tumor measurement within 4 weeks (28 days) prior to enrollment.

  * Chest: CT scan with intravenous contrast if the contrast is not medically contraindicated.
  * Abdomen: CT scan with intravenous and oral contrast if the contrast is not medically contraindicated.
  * Pelvis: CT scan with intravenous and oral contrast if the contrast is not medically contraindicated.
  * Brain: CT scan or MRI
  * Bone: Whole body Bone Scintigraphy or PET scan
* Female 18 years of age or older at the time the written informed consent is obtained.
* ECOG Performance Status of 0 or 1.
* Adequate organ and hematological function as evidenced by the following laboratory studies within 2 weeks (14 days) of study enrollment, unless stated otherwise:

  * Cardiac function, as follows:

    * Normal sinus rhythm (no significant ECG changes)
    * Left ventricular ejection fraction ≥ Lower Limit of Normal, as determined by echocardiogram or MUGA scan, according to institutional standards within 28 days prior to study enrollment.
  * Hematological function, as follows:

    * Absolute neutrophil count ≥ 1.5 x 109/L
    * Platelet count ≥ 100 x 109/L and ≤ 850 x 109/L
    * Hemoglobin ≥ 9 g/dL.
    * PTT and INR < 1.5 x ULN.
  * Renal function, as follows:

    * Serum creatinine ≤ 175 µmol/L (= 2mg/dL). If creatinine is between 140-175 µmol/L, creatinine clearance (calculated or measured) should be > 40 mL/min.
    * Urinary protein quantitative value of ≤ 30 mg/dL in urinalysis or ≤ 1 + on dipstick unless protein is < 500 mg in a 24-hour urine sample.
  * Hepatic function, as follows:

    * Aspartate aminotransferase (AST) ≤ 2.5 x ULN
    * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Total bilirubin ≤ 1 x ULN
* Patients of child-bearing potential and sexually active must provide a negative pregnancy test within 7 days prior to enrollment.
* More than 4 weeks since prior therapy for breast cancer
* No other concurrent investigational or commercial agents or therapies for metastatic breast cancer
* No prior capecitabine or fluorouracil for metastatic breast cancer
* More than 4 weeks since prior radiotherapy **Previously irradiated area(s) must not be the only site of disease**
* More than 4 weeks since prior major surgery

Exclusion Criteria:

Disease Related:

* Current or prior history of central nervous system metastasis.
* Common Terminology Criteria for Adverse Events (CTCAE) v. 3.0 peripheral neuropathy ≥ grade 2 at enrollment.
* Average systolic blood pressure > 150 mm Hg or average diastolic blood pressure > 90 mm Hg (average blood pressure of the 3 separate blood pressure values measured according to the Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure.
* History of arterial or venous thrombosis within 1 year prior to enrollment.
* History of bleeding diathesis or bleeding within 14 days of enrollment.
* Major surgical procedure within 4 weeks (28 days) prior to enrollment.
* Minor surgical procedure, placement of access device, or fine needle aspiration within 7 days of enrollment.
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or malignancy (other than in situ cervical cancer, or basal cell cancer of the skin), unless treated with curative intent and without evidence of disease for ≥ 3 years before study enrollment.
* Clinically significant cardiac disease within 12 months of study enrollment, including myocardial infarction, unstable angina, grade II or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or ongoing arrhythmias requiring medication or pacemaker.
* Non-healing wound, ulcer or fracture.
* Ongoing or active infection.
* Known chronic hepatitis.

Medications:

* Currently or previously treated with small molecule inhibitors of VEGF including, but not limited to, SU11248 (sunitinib), PTK787 (vatalinib), AZD 2171, AZD 6474, AEE-788, BAY 43-9006 (sorafenib) and motesanib.
* Treatment with rifampin, carbamazepine, rifabutin or phenobarbital within 14 days prior to study enrollment.
* Treatment with strong CYP 3A inhibitors or inducers such as ketoconazole, itraconazole, fluconazole, clarithromycin, erythromycin, nefazodone, or any HIV protease inhibitors within 7 days prior to study enrollment.
* Treatment with immune modulators such as cyclosporine and tacrolimus within 7 days prior to study enrollment.
* Treatment with herbal medications containing St. John's Wort within 7 days prior to study enrollment.
* Concomitant therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMS), given for breast cancer prevention or for osteoporosis. Patients must have discontinued these agents prior to enrollment.

General:

* Known hypersensitivity to any study medications (motesanib, and Chinese Hamster Ovary cell products or other human or humanized recombinant proteins) or Cremaphor.
* Any condition which in the investigator's opinion makes the patient unsuitable for the study participation. This includes substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Participation in other investigational device drug trials, or administration of other investigational treatments within 30 days prior to study enrollment.
* Pregnant (i.e., positive beta-human chorionic gonadotropin test)
* Not willing to use a highly effective method of birth control (i.e. those which result in low failure rates, less than 1% per year), such as nonhormonal IUD, condoms, sexual abstinence or vasectomised partner.

**Contraception must be used during the study and for 6 months after last dose of study treatment**

* Unable to swallow oral medications.
* Inability to comply with protocol and/or not available for follow-up assessments.
* Males of any age.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Up to 3 years or disease progression
  Progression-free survival (PFS) is defined as the time from the date of enrollment to the first occurrence of having documented disease progression or death due to any cause. Evaluation of target lesions and non-target lesions will be in accordance with the RECIST criteria.
  During the study, assessments of tumor response will take place every 6 weeks. Confirmation of objective response, when applicable, must be performed at a minimum of 4 weeks after the first response has been recorded.

SECONDARY OUTCOMES:
Maximum Tolerated Dose of Motesanib | 120 days
  Maximum tolerated dose (MTD) of Motesanib to be determined in the first 3-6 patients enrolled to study (Phase I portion).
Overall Response Rate | Through 28 days post-treatment
  The best overall response in an individual patient according to the RECIST criteria is the best response recorded from the time of study entry till disease progression/recurrence. The patient's overall best response can be complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD).
  Patients with CR or PR are deemed as responders. Patients with no tumor assessment after the study entry are to be considered as non-responders.
Toxicity | Through 28 days post-treatment
  To determine the toxicity of motesanib, ixabepilone, and capecitabine, using a single arm design trial.
Correlation of Tumor Levels | Up to 3 years or disease progression
  To correlate quantitative tumor levels of motesanib-relevant markers PDGFR, VEGFR, C-Kit, and their ligands with response, survival, and time to disease progression in patients treated on this regimen.
Pharmacokinetics of Study Regimen | Through 28 days post-treatment
  To investigate the pharmacokinetics of motesanib (Cmin), ixabepilone (concentration at the end of infusion), and capecitabine in the combination therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Mitchell, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/